CLINICAL TRIAL: NCT06121089
Title: Study of the Oncological Outcomes of Ileocecal Resection With D3 for Cecal Cancer
Brief Title: Local Cecal Cancer - Optimization of Surgical Treatment
Acronym: LoCCOSTe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2022
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Colonic Neoplasms Malignant; Cecal Neoplasms
Keywords: Colorectal cancer; Segmental colonic resection; Ileocecal resection; Cecal cancer; Right hemicolectomy
MeSH Terms: conditions — Cecal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will be randomly divided into two groups in a 1:1 ratio.
  1. Research group (ICR) - Laparoscopy ileocecal resection with extended D3 lymphadenectomy (including 201, 202, 203 and 213 groups of lymph nodes). The minimum distance from the tumor is 10 cm, along the line of adequate blood supply. Next step - formation of a manual double-row ileo-ascendo-anastomosis.
  2. Control group (RHC) - Laparoscopy right hemicolectomy with D3 lymphadenectomy (including 211, 212, 221, 222-rt groups of lymph nodes). Next step - formation of a manual double-row ileo-transverse-anastomosis.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopy ileocecal resection with extended D3 lymphadenectomy. (Active Comparator): Ileocecal resection with extended D3 lymphadenectomy.
  Interventions: Procedure: ileocecal resection with extended D3 lymphadenectomy.
- Laparoscopy right hemicolectomy with D3 lymphadenectomy. (Experimental): Right hemicolectomy with D3 lymphadenectomy
  Interventions: Procedure: Right hemicolectomy with D3 lymphadenectomy.

INTERVENTIONS:
Procedure: ileocecal resection with extended D3 lymphadenectomy. — Laparoscopy ileocecal resectionith extended D3 lymphadenectomy including 201, 202, 203 and 213 groups of lymph nodes. Manual double-row ileo-ascendo-anastomosis.
  Arms: Laparoscopy ileocecal resection with extended D3 lymphadenectomy.
Procedure: Right hemicolectomy with D3 lymphadenectomy. — Laparoscopy right hemicolectomy with D3 lymphadenectomy including 201, 202, 203, 213, 211, 212, 221, 222-rt groups of lymph nodes. Manual double-row ileo-transverse-anastomosis.
  Arms: Laparoscopy right hemicolectomy with D3 lymphadenectomy.

SUMMARY:
The purpose of this study is to determine the clinical efficacy, safety, and oncologic outcomes of ileocecal resection (ICR) with D3 lymphadenectomy compared to standard right hemicolectomy(RHC) for cecal cancer.

DETAILED DESCRIPTION:
The design involves random allocation of eligible patients to ICR or RHC group in 1:1 ratio.

Requirements applied to centers participating in the trial and surgeons performing procedures are described in the protocol and refer to center volume and surgeon's experience.

Regular quality control includes the requirement to photograph the surgical specimen with a mark to determine the extent of lymphadenectomy performed and the number of the lymph node group.

After surgery patients are treated according to local standards, regardless of whether ICR or RHC was performed. Short-term and long-term outcomes are recorded according to the protocol.

Intervention. In all cases the tumor is localized in the area of the cecum; the border of the transition to the ascending colon is the upper lip of the ileocecal valve. The patient is not included in the study if the preoperative stage of examination reveals: synchronous cancer, distant metastasis (M1), locally advanced nature of the primary tumor (cT > 3).

All patients will be randomly divided into two groups in a 1:1 ratio.

1. Research group (ICR) - Laparoscopy ileocecal resection with extended D3 lymphadenectomy (including 201, 202, 203 and 213 groups of lymph nodes). The minimum distance from the tumor is 10 cm, along the line of adequate blood supply. Next step - formation of a manual double-row ileo-ascendo-anastomosis.
2. Control group (RHC) - Laparoscopy right hemicolectomy with D3 lymphadenectomy (including 211, 212, 221, 222-rt groups of lymph nodes). Next step - formation of a manual double-row ileo-transverse-anastomosis.

Expected Results. The ICR will improve the short-term results of treatment of patients with cecal cancer compared with the standard RHC technique without affecting long-term results.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* ECOG status 0-2.
* Histologically confirmed adenocarcinoma of the colon.
* Clinical stage T1-3; N+; M0.
* The physical status from ASA classification I, II, III or IV.
* Written informed consent.

Exclusion Criteria:

* Synchronous or metachronous malignancy.
* Locally-advanced tumor (T>3).
* Presence of distant metastases (M1).
* Complicated tumor: obstruction, perforation.
* Neoadjuvant chemotherapy.
* Medical contraindications for surgical treatment.
* Pregnancy or breast feeding.
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival. | 5 years after the last patient.
  Overall survival of patients.
Disease-free survival. | 3 years after the last patient.
  Survival without local or distant recurrence.
Disease-free survival. | 5 years after the last patient.
  Survival without local or distant recurrence.

SECONDARY OUTCOMES:
Postoperative morbidity. | The first 30 days after surgery.
  Complications after surgery.
Postoperative mortality. | The first 30 days after surgery.
  Death after surgery.
Total number of lymph nodes removed. | Post-intervention at week 3.
  Number of removed lymph nodes according to pathomorphological evaluation.
Total number of metastatic lymph nodes and correlation by group. | Post-intervention at week 3.
  The ratio of affected lymph nodes into groups (201, 202, 203, 213, 211, 212, 221 or 222-rt) depending on the type of surgical treatment. Based on pathological assessment.
Total length of removed bowel. | Post-intervention at week 3.
  Average length of removed bowel in both groups according to pathomorphological evaluation (millimeters).
Area of mesentery removed. | Post-intervention at week 3.
  Average area of the removed mesentery in each groups according to pathomorphological evaluation (square centimetre - sq.cm).
Description of blood loss during the intraoperative period. | During the surgery.
  Average blood loss during surgery in each group (ml).
Operation time. | Immediately after the surgery.
  Average operation time for each group (minutes - min).
Conversion. | During the surgery.
  The total number of conversions for each group.
Number of days of inpatient treatment. | During hospitalization up to 4 weeks
  Average number of days of inpatient treatment.

OTHER OUTCOMES:
Determination of the number and level of lymph node involvement. | Period of examination before surgery.
  X-ray assessment (Node-RADS classification) of clinical stage (N0 or N+) and distribution of suspicious lymph nodes into groups.
Quality of life in patients after ICR and RHC using questionnaire. | 30 days post-surgery.
  Questionnaires by European Organization for Research and Treatment of Cancer. EORTC QLQ - CR29.

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow Clinical Scientific Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
We are not planning to share personal patient data.